CLINICAL TRIAL: NCT05714085
Title: A Phase 2/3 Randomized, Placebo-Controlled, Double-blind, Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Vericiguat in Pediatric Participants With Heart Failure Due to Systemic Left Ventricular Systolic Dysfunction (VALOR)
Brief Title: Efficacy, Safety, and Pharmacokinetics of Vericiguat in Pediatric Participants With Heart Failure Due to Left Ventricular Systolic Dysfunction (MK-1242-036)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1242-036; MK-1242-036 (Other: MSD); 2022-501238-52-00 (Registry Identifier: EU CT); U1111-1275-1768 (Registry Identifier: UTN); MK-1242-043 (Other: MSD Obsolete Identifier); 2021-004399-33 (EudraCT Number); NCT06428383 (obsolete NCT alias)
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure; Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left | interventions — vericiguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Base Period: Vericiguat (Experimental): Participants in the Base Period receive 2.5 mg or 5 mg or 10 mg vericiguat administered orally once daily in tablet form for 52 weeks; or 0.2 mg/mL or 1 mg/mL vericiguat administered orally once daily in suspension form for 52 weeks.
  Interventions: Drug: Vericiguat tablet; Drug: Vericiguat suspension
- Base Period: Placebo (Placebo Comparator): Participants in the Base Period receive placebo for vericiguat administered orally once daily in tablet form for 52 weeks, or administered orally once daily in suspension form for 52 weeks.
  Interventions: Drug: Placebo tablet; Drug: Placebo suspension
- Extension Period: Vericiguat (Experimental): Participants in the Extension Period receive either 2.5 mg or 5 mg or 10 mg vericiguat administered orally once daily in tablet form; or 0.2 mg/mL or 1 mg/mL vericiguat administered orally once daily in suspension form; following completion of the Base Period.
  Interventions: Drug: Vericiguat tablet; Drug: Vericiguat suspension

INTERVENTIONS:
Drug: Vericiguat tablet — 2.5 mg or 5 mg or 10 mg vericiguat administered orally once daily in tablet form
  Other Names: MK-1242
  Arms: Base Period: Vericiguat; Extension Period: Vericiguat
Drug: Vericiguat suspension — 0.2 mg/mL or 1 mg/mL vericiguat administered orally once daily in suspension form
  Other Names: MK-1242
  Arms: Base Period: Vericiguat; Extension Period: Vericiguat
Drug: Placebo tablet — Placebo for vericiguat administered orally once daily in tablet form
  Other Names: Placebo for MK-1242
  Arms: Base Period: Placebo
Drug: Placebo suspension — Placebo for vericiguat administered orally once daily in suspension form
  Other Names: Placebo for MK-1242
  Arms: Base Period: Placebo

SUMMARY:
This study aims to compare the efficacy of vericiguat versus placebo on change in n-terminal pro-brain natriuretic peptide (NTproBNP) from baseline to Week 16 of the Base Period. The primary hypothesis is that vericiguat is superior to placebo in reducing NT-proBNP at Week 16 of the Base Period.

DETAILED DESCRIPTION:
As of Protocol Amendment 2, the separate open-label extension arm of study MK-1242-043 (NCT06428383) will be incorporated into the present MK-1242-036 study as an extension period. Participants from the Base Period will be provided the opportunity to participate in the optional open-label Extension Period if eligible. After all ongoing participants are transferred into the extension period of MK-1242-036, MK-1242-043 (NCT06428383) will be formally closed.

ELIGIBILITY:
Inclusion Criteria:

* Has symptomatic chronic heart failure (HF) resulting from systemic left ventricular (LV) systolic dysfunction.
* Has biventricular physiology with a morphologic systemic left ventricle.
* Is currently receiving stable medical therapy for HF.
* Has left ventricular ejection fraction (LVEF) <45% assessed within 3 months before randomization.
* Is of any sex/gender, from >28 days to <18 years of age inclusive. Must weigh ≥3 kg to participate.
* Female is eligible to participate if not pregnant or breastfeeding, and at least one of the following: is not a participant of childbearing potential (POCBP); or is a POCBP who uses a highly effective contraceptive method; has a negative highly sensitive pregnancy test; abstains from breastfeeding during the study intervention period and for at least 30 days after study intervention; and their medical history; their menstrual history, and recent sexual activity has been reviewed.
* Extension Period: Was randomized, received at least 1 dose of study intervention (vericiguat or placebo), did not permanently discontinue study intervention, and completed the Week 52 visit and safety follow-up period of the Base Period

Exclusion Criteria:

* Is clinically unstable-with at least one of the following: has symptomatic hypotension or is hypotensive for age, recent use of intravenous (IV) inotrope and/or IV vasodilator, or recent IV diuretic.
* Has a known allergy or sensitivity to vericiguat, any of its constituents, or any other soluble guanylate cyclase (sGC) stimulator.
* Has a history of single ventricle heart disease or has a morphologic systemic right ventricle.
* Has undergone heart transplantation, is awaiting heart transplantation United Network for Organ Sharing (UNOS) Class 1A or equivalent, is receiving continuous IV infusion of an inotrope, or has an implanted ventricular assist device.
* Has sustained or symptomatic dysrhythmia uncontrolled with drug or device therapy.
* Has had recent cardiovascular (CV) surgical procedure or percutaneous intervention to palliate or correct congenital CV malformations.
* Has unoperated or residual hemodynamically significant congenital cardiac malformations.
* Has hypertrophic or restrictive cardiomyopathy.
* Has active myocarditis or has been recently diagnosed with presumed or definitive myocarditis.
* Has acute coronary syndrome, undergone recent coronary intervention, or indication for coronary revascularization.
* Has symptomatic carotid stenosis or other symptomatic cerebrovascular disease
* Has severe pulmonary hypertension.
* Requires continuous home oxygen for significant pulmonary disease and/or has known interstitial lung disease.
* Has severe chronic kidney disease.
* Has hepatic disorder such as hepatic encephalopathy, hepatic laboratory abnormalities or Child Pugh Class C.
* Has a gastrointestinal or biliary disorder that could impair absorption, metabolism, or excretion of medications.
* Has significant bone disease (other than osteopenia) that in the assessment of the investigator can alter bone formation
* Has concurrent or anticipated concomitant use of phosphodiesterase type 5 inhibitors or an sGC stimulator.
* Has received a COVID-19 vaccination within 1 week before randomization.

Ages: 29 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 342 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2032-04-15 (Estimated); Study Completion 2032-04-15 (Estimated)

PRIMARY OUTCOMES:
Base Period: Change from baseline to Week 16 in N-terminal pro-brain natriuretic peptide (NT-proBNP) | Baseline and Week 16 of Base Period
  The change from baseline to Week 16 of the Base Period in log-transformed NT-proBNP will be reported.
Extension Period: Percentage of participants with one or more adverse events (AEs) | Includes data collected up to a maximum of approximately 8 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with one or more AEs in the Extension Period will be reported.
Extension Period: Percentage of participants who discontinued study drug due to an AE | Includes data collected up to a maximum of approximately 8 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study drug in the Extension Period due to an AE will be reported.

SECONDARY OUTCOMES:
Base Period: Change from baseline to Week 52 in log-transformed NT-proBNP | Baseline and Week 52 of Base Period
  The change from baseline to Week 52 of the Base Period in log-transformed NT-proBNP will be reported.
Base Period: First event of cardiovascular (CV) death, heart failure hospitalization (HFH), or worsening of heart failure (HF) without hospitalization | Up to Week 54 of Base Period
  The time from randomization to the first event of CV death, HFH, or worsening of HF without hospitalization will be reported for the Base Period.
Base Period: Percentage of participants with one or more adverse events (AEs) | Up to Week 54 of Base Period
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with one or more AEs in the Base Period will be reported.
Base Period: Percentage of participants who discontinued study drug due to an AE | Up to Week 52 of Base Period
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study drug in the Base Period due to an AE will be reported.
Base Period: Area under the curve from time 0-24 hours post-dose (AUC0-24) of plasma vericiguat | Pre-dose, 2, 6, 16, 32 and 52 weeks post-dose (Base Period)
  Blood samples were collected at pre-specified time points pre- and post-dose and used to estimate the area under the curve from time 0-24 hours post-dose (AUC0-24) of plasma vericiguat.
Base Period: Half-life (t1/2) of vericiguat in plasma | Pre-dose, 2, 6, 16, 32 and 52 weeks post-dose (Base Period)
  Blood samples were collected at pre-specified time points pre- and post-dose and used to estimate the t1/2 of vericiguat in plasma.
Base Period: Oral clearance (CL/F) of plasma vericiguat | Pre-dose, 2, 6, 16, 32 and 52 weeks post-dose (Base Period)
  Blood samples were collected at pre-specified time points pre- and post-dose and used to estimate the CL/F of vericiguat in plasma.
Extension Period: Change from extension period baseline to extension period Week 16 in NT-proBNP | Extension Period Baseline (Study Week 54) and Extension Period Week 16 (Study Week 70)
  The change from the Extension Period baseline to Week 16 of the Extension Period in log-transformed NT-proBNP will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (97):
- United States (18):
  - Loma Linda University Health System ( Site 0008), Loma Linda, California
  - The Regents of the University of California - Los Angeles (UCLA Pediatrics) ( Site 0002), Los Angeles, California
  - Children's Hospital Colorado ( Site 0012), Aurora, Colorado
  - Children's National Medical Center ( Site 0020), Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital ( Site 0029), St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Arthur M. Blank Hospital ( Site 0001), Atlanta, Georgia
  - Boston Children's Hospital ( Site 0035), Boston, Massachusetts
  - C.S. Mott Children's Hospital ( Site 0033), Ann Arbor, Michigan
  - Washington University-Pediatric Cardiology/ St. Louis Children's Hospital ( Site 0006), St Louis, Missouri
  - Columbia University Medical Center-Pediatric Cardiology ( Site 0016), New York, New York
  - The Children's Hospital at Montefiore ( Site 0030), The Bronx, New York
  - Cincinnati Children's Hospital Medical Center ( Site 0034), Cincinnati, Ohio
  - Cleveland Clinic-Cleveland Clinic Chidren's ( Site 0022), Cleveland, Ohio
  - Children's Hospital of Philadelphia (CHOP) ( Site 0004), Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh ( Site 0010), Pittsburgh, Pennsylvania
  - Le Bonheur Children's Hospital ( Site 0007), Memphis, Tennessee
  - Children's Health-The Heart Center ( Site 0015), Dallas, Texas
  - Seattle Children's Hospital-Cardiology/Fetal Therapy ( Site 0019), Seattle, Washington
- Belgium (3):
  - Centre Hospitalier Régional de la Citadelle ( Site 0302), Liège, Liege
  - UZ Gent ( Site 0301), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0300), Leuven, Vlaams-Brabant
- Brazil (2):
  - Instituto Dante Pazzanese de Cardiology ( Site 0402), São Paulo, São Paulo
  - Incor - Instituto do Coracao ( Site 0400), São Paulo
- Canada (2):
  - Stollery Children's Hospital ( Site 0501), Edmonton, Alberta
  - Centre intégré universitaire de santé et de services sociaux-Centre de recherche du CHUS ( Site 0502), Sherbrooke, Quebec
- Colombia (5):
  - Clinica Somer ( Site 0607), Rionegro, Antioquia
  - Ciensalud Ips S A S ( Site 0608), Barranquilla, Atlántico
  - Fundación Cardioinfantil Instituto de Cardiología ( Site 0603), Bogotá, Bogota D.C.
  - Fundación Valle del Lili ( Site 0604), Cali, Valle del Cauca Department
  - Clínica Imbanaco S.A.S ( Site 0602), Cali, Valle del Cauca Department
- Rigshospitalet-BørneUngeAfdelingen ( Site 0800), Copenhagen, Capital Region, Denmark
- Tampereen yliopistollinen sairaala-Pediatric Early Phase Trials Unit ( Site 0900), Tampere, Pirkanmaa, Finland
- France (6):
  - CHU Bordeaux Haut-Leveque ( Site 1000), Pessac, Aquitaine
  - CHU Lille - Institut Coeur Poumon ( Site 1005), Lille, Nord
  - Centre Hospitalier Universitaire de Nantes - Hôpital Femme-Enfant-Adolescent Chu De Nantes ( Site 1002), Nantes, Pays de la Loire Region
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone ( Site 1003), Marseille, Provence-Alpes-Côte d'Azur Region
  - Hôpital Universitaire Necker Enfants Malades ( Site 1001), Paris
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - Centre Hospitalo Universita ( Site 1004), Paris
- Germany (5):
  - Universitaetsklinikum Freiburg ( Site 1102), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Heidelberg ( Site 1100), Heidelberg, Baden-Wurttemberg
  - Kinderklinik des Uni-Klinikums Erlangen ( Site 1104), Erlangen, Bavaria
  - Medizinische Hochschule Hannover ( Site 1108), Hanover, Lower Saxony
  - Deutsches Herzzentrum Berlin ( Site 1101), Berlin
- Gottsegen György Országos Kardiovaszkuláris Intézet-Gyermeksziv Kozpont ( Site 1300), Budapest, Hungary
- Children's Health Ireland (CHI) at Crumlin ( Site 1400), Dublin, Ireland
- Italy (4):
  - IRCCS Istituto Giannina Gaslini ( Site 1603), Genoa, Liguria
  - Ospedale Pediatrico Bambino Gesù IRCCS ( Site 1602), Rome, Roma
  - A.O.Universitaria Meyer ( Site 1600), Florence, Tuscany
  - Azienda Ospedale - Università Padova ( Site 1601), Padua, Veneto
- Malaysia (5):
  - Hospital Universiti Sains Malaysia ( Site 1703), Kota Bharu, Kelantan
  - University Malaya Medical Centre ( Site 1701), Lembah Pantai, Kuala Lumpur
  - Hospital Queen Elizabeth II ( Site 1706), Kota Kinabalu, Sabah
  - Hospital Tunku Azizah-Paediatric ( Site 1700), Kuala Lumpur
  - Institut Jantung Negara ( Site 1705), Kuala Lumpur
- Mexico (8):
  - Morales Vargas Centro de Investigacion ( Site 1810), León, Guanajuato
  - CINVEC Medica ( Site 1814), Guadalajara, Jalisco
  - Instituto Nacional de Pediatria ( Site 1803), Mexico City, Mexico City
  - INVECORDIS S.C. ( Site 1808), Hacienda de Las Palmas, State of Mexico
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares ( Site 1800), Ciudad Madero, Tamaulipas
  - Centro de Atención e Investigación Clínica ( Site 1813), Aguascalientes
  - UROLAP ( Site 1812), Colima
  - Instituto Nacional de Cardiologia Ignacio Chavez ( Site 1804), México
- Netherlands (3):
  - Erasmus Medisch Centrum ( Site 1900), Rotterdam, South Holland
  - University Medical Center Groningen ( Site 1901), Groningen
  - Universitair Medisch Centrum Utrecht ( Site 1902), Utrecht
- Auckland City Hospital ( Site 2000), Auckland, New Zealand
- Instituto Nacional Cardiovascular INCOR Carlos Peschiera Carrillo - EsSalud ( Site 2100), Jesús María, Lima, Peru
- Uniwersyteckie Centrum Kliniczne-Klinika Kardiologii Dziecięcej i Wad Wrodzonych Serca ( Site 2302), Gdansk, Pomeranian Voivodeship, Poland
- Portugal (3):
  - Unidade Local de Saude Lisboa Ocidental - Hospital de Santa Cruz ( Site 2401), Lisbon, Lisbon District
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 2402), Lisbon
  - Unidade Local de Saúde de São João ( Site 2403), Porto
- Singapore (2):
  - National University Hospital-Paediatrics ( Site 2600), Singapore, South West
  - KK Women's and Children's Hospital ( Site 2601), Singapore, South West
- South Africa (2):
  - TREAD Research ( Site 2700), Cape Town, Western Cape
  - Children's Heart Disease Research Unit ( Site 2704), Cape Town, Western Cape
- South Korea (4):
  - Pusan National University Yangsan Hospital ( Site 2802), Pusan, Kyongsangnam-do
  - Seoul National University Hospital ( Site 2803), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 2800), Seoul
  - Samsung Medical Center ( Site 2801), Seoul
- Spain (6):
  - Hospital Sant Joan de Déu-Pediatric cardiology ( Site 2902), Esplugues de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 2903), Barcelona, Catalonia
  - Hospital Materno-Infantil Teresa Herrera ( Site 2905), A Coruña, La Coruna
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON ( Site 2904), Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz ( Site 2912), Madrid
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO ( Site 2907), Seville
- Sweden (2):
  - Skånes Universitetssjukhus Lund ( Site 3000), Lund, Skåne County
  - Astrid Lindgrens Barnsjukhus ( Site 3001), Stockholm, Stockholm County
- Thailand (3):
  - Faculty of Medicine Siriraj Hospital ( Site 3200), Bangkok, Bangkok
  - Faculty of Medicine - Khon Kaen University ( Site 3202), Muang, Changwat Khon Kaen
  - Maharaj Nakorn Chiang Mai Hospital-Department of Pediatrics ( Site 3201), Chiang Mai
- Turkey (Türkiye) (5):
  - Hacettepe Universite Hastaneleri ( Site 3304), Ankara
  - Baskent Universitesi Ankara Hastanesi ( Site 3301), Ankara
  - Ankara Bilkent Şehir Hastanesi. ( Site 3300), Ankara
  - Dr. Siyami Ersek Göğüs Kalp Ve Damar Cerrahisi Eğitim Ve Araştırma Hastanesi ( Site 3302), Istanbul
  - S.B.Ü. DR. BEHÇET UZ ÇOCUK HASTALIKLARI VE CERRAHİSİ EĞİTİM VE ARAŞTIRMA HASTANESİ ( Site 3303), Izmir
- United Kingdom (2):
  - Great Ormond Street Hospital For Children NHS Foundation Trust ( Site 3401), London, London, City of
  - Freeman Hospital ( Site 3400), Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Fritsch A, Meyer M, Blaustein RO, Trujillo ME, Kauh E, Roessig L, Boettcher M, Becker C. Clinical Pharmacokinetic and Pharmacodynamic Profile of Vericiguat. Clin Pharmacokinet. 2024 Jun;63(6):751-771. doi: 10.1007/s40262-024-01384-1. Epub 2024 Jun 25. PMID 38916717
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26221&tenant=MT_MSD_9011
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/